CLINICAL TRIAL: NCT02147418
Title: An Observational, Single-Institution Pilot/Feasibility Study of Exosome Testing as a Screening Modality for Human Papillomavirus-Positive Oropharyngeal Squamous Cell Carcinoma
Brief Title: Exosome Testing as a Screening Modality for Human Papillomavirus-Positive Oropharyngeal Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 1310
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Oropharyngeal Cancer
Keywords: Head and neck cancer; Throat cancer; Human papillomavirus; HPV; Exosome; Diagnostic; Early Detection
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All oropharyngeal rinse (gargle) specimens will be processed within 24 hours of collection. Any remaining material after testing will be stored for a period not to exceed 1 year in a secure location.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: HPV-positive Cancer: Oropharyngeal cancer patients testing positive for human papillomavirus (HPV)
- Group 2: HPV-positive Cancer: Oropharyngeal cancer patients who test positive for human papillomavirus (HPV)
- Group 3: Healthy Controls: Patients with benign conditions

SUMMARY:
Cancer of the oropharynx (middle, side and back walls of the throat; back of the tongue; soft palate, and tonsils), or oropharyngeal squamous cell carcinoma (OPSCC), has been on the rise in the United States. Human papillomavirus (HPV) has been recognized in many of these cancers, and testing for HPV has contributed to the higher reported rates of OPSCC. In this study, our goal is to develop a new test that can detect certain HPV proteins in the blood or saliva to help improve detection of OPSCC.

DETAILED DESCRIPTION:
While secondary screening strategies have successfully reduced the rate of HPV-positive cervical cancers, an effective screening modality for HPV-OPSCC does not exist. A central problem in the early diagnosis of HPV-OPSCC is the relative inaccessibility of the tonsillar crypts, where oncogenic infections are thought to originate. Unlike the relatively smooth surface of the cervix which permits mechanical sampling with Pap tests and which can be evaluated visually for evidence of dysplasia, much of the tonsillar epithelium is found below the surface in a complex network. As a consequence, any screening modality cannot depend upon direct access to malignant lesions. What is needed is a minimally invasive, diffusible or circulating marker of HPV-OPSCC, and a means to collect and detect it.

ELIGIBILITY:
Inclusion Criteria (Cancer Patients):

* Male or Female
* Age greater than or equal to 18
* Previously untreated, pathologically confirmed OPSCC (HPV+ or HPV-)
* Ability to understand study information and provide written consent for participation.

Inclusion Criteria (Non-cancer Patients):

* Male or Female
* Age greater than or equal to 18
* Ability to understand study information and provide written consent for participation

Exclusion Criteria:

* Age less than 18 years
* Prisoners
* Pregnant women
* Patients with mental disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population will consist of adults presenting to the Division of Otolaryngology - Head and Neck Surgery at the University of New Mexico with previously untreated OPSCC. Both HPV-positive and HPV-negative malignancies will be collected as the study and control groups, respectively. In addition, saliva samples will be collected from patients presenting with benign conditions as a further negative control.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Cultured Cell Exosome Protein Signature Outcome Measure | 1 month
  The presence of unique proteins obtained from primary cell cultures derived from HPV-OPSCC confirmed patients will be compared to normal tonsillar epithelial cells and established cell lines. The distribution of these protein signatures will be compared in HPV-OPSCC and normal epithelial cells.

OTHER OUTCOMES:
Exosome Signatures Oropharyngeal Rinse Measure | 1 month
  Compare exosome protein signatures generated from cells obtained through oropharyngeal rinses of patients with HPV-positive OPSCC and normal controls to identify an exosome protein marker that is absent (or present at a different, statistically significant level) in the oropharyngeal rinses of normal controls.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cowan, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Cancer Center — http://cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org